CLINICAL TRIAL: NCT06832202
Title: A Phase II Study of HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination With Trastuzumab Deruxtecan (T-DXd) in HER2-low, Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer Patients With Intolerable Adverse Reaction or Disease Progression on Standard of Care
Brief Title: A Phase II Study of HLX22 in Combination With Trastuzumab Deruxtecan in HER2-low, Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX22-BC201
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-01

CONDITIONS: HER2-low Hormone Receptor Positive Breast Cancer
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): HLX22(15 mg/kg) + Trastuzumab Deruxtecan( 5.4 mg/kg), Q3W
  Interventions: Drug: HLX22; Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: HLX22 — HLX22 15mg/kg Q3W
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan 5.4mg/kg Q3W

SUMMARY:
This is a Phase II Study of HLX22 in Combination with Trastuzumab Deruxtecan (T-DXd) in HER2-low, Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer Patients with Disease Progression or Intolerable Adverse Reaction on Standard of Care. Eligible subjects will be treated with the study drug until the loss of clinical benefit, death, intolerable toxicity, withdrawal of informed consent, or other reasons specified by the protocol (whichever occurs first).

DETAILED DESCRIPTION:
experimental group: HLX22(15 mg/kg) + Trastuzumab Deruxtecan( 5.4 mg/kg), once every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female who are at least 18 years of age on the day of signing the informed consent.
2. With histologically confirmed diagnosis of HER2-low, Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer.
3. HER2-low defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested) as assessed by a central laboratory on metastatic tumor and was never previously HER2-positive，and was documented HR+ disease in the metastatic setting
4. Had measurable disease according to the RECIST v1.1, the target lesion must not be a bone metastatic lesion only.
5. ECOG PS: 0-1.
6. Expected survival ≥ 6 months.
7. Had adequate organ function

Exclusion Criteria:

1. Patients with other malignant tumors within 3 years before the randomization
2. Previous treatment with any HER2-target therapy
3. Uncontrolled or significant cardiovascular disease or infection
4. Lung-specific intercurrent clinically significant illnesses
5. Prior documented interstitial lung disease (ILD)/ pneumonitis that required steroids, current ILD/ pneumonitis, or suspected ILD/ pneumonitis
6. Patients with spinal cord compression or clinically active central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years
  Progression-Free Survival (PFS) assessed by IRRC (Independent Radiology Review Committee) per RECIST 1.1 . PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.
Objective response rate (ORR) | Up to 2 years
  Objective Response Rate (ORR) assessed by IRRC per RECIST v1.1. ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1

SECONDARY OUTCOMES:
PFS | Up to 5 years
  PFS assessed by investigator per RECIST 1.1 . PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.
ORR | Up to 2 years
  ORR assessed by investigator per RECIST v1.1. ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1
Aderse events (AE) | Up to 5 years
  AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China